CLINICAL TRIAL: NCT03679260
Title: Carbohydrate and Prostate Study 3: Carbohydrate Restricted Diet Intervention for Men on Prostate Cancer Active Surveillance
Brief Title: Carbohydrate Restricted Diet Intervention for Men on Prostate Cancer Active Surveillance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Freedland, Director, Center for Integrated Research in Cancer and Lifestyle; Co-Director, Cancer Genetics and Prevention Program; Professor, Surgery, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT2018-06-FREEDLAND-AS3
Record Dates: First submitted 2018-09-11; First posted 2018-09-20 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate Adenocarcinoma; Active Surveillance; Diet; Weight Loss; low carb; Ketogenic Diet; Ketogenic
MeSH Terms: conditions — Prostatic Neoplasms; Weight Loss | interventions — Diet, Carbohydrate-Restricted; Nutritionists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Carbohydrate restricted diet and phone counseling with dietitian. After 6 months, patients will crossover to a non-restricted diet.
  Interventions: Other: Carbohydrate restricted diet; Other: Non-restricted diet; Other: Phone counseling with dietitian
- Arm B (Experimental): Non-restricted diet and after 6 months, patients will crossover to a carbohydrate restricted diet and phone counseling with dietitian
  Interventions: Other: Carbohydrate restricted diet; Other: Non-restricted diet; Other: Phone counseling with dietitian

INTERVENTIONS:
Other: Carbohydrate restricted diet — 20 grams total carbs/day
Other: Non-restricted diet — Subject follows normal diet
Other: Phone counseling with dietitian — Weekly calls with dietitian

SUMMARY:
This phase 2 waitlist-controlled, randomized trial is designed to compare the difference in proliferative index (Ki67) between carbohydrate restricted diet and usual care over a 6 month period in men with prostate cancer who have been placed on Active Surveillance. Eligible patients include men over 18 years old, BMI >25, with their most recently performed biopsy pathologically confirming prostate adenocarcinoma who have been placed on AS. Arms of the trial will be randomized 1:1 in a crossover approach, with Arm A receiving a carb restricted diet over 6 months then SOC and Arm B receiving the waitlist control arm (i.e. SOC then allowed to go on diet after 6 months). Ki67 will be performed on tissue from the most recent biopsy at the beginning of the study and again on tissue obtained in the 6 month SOC biopsy. Every patient will be on the study for 12 months, and the study will continue for approximately 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed prostate adenocarcinoma
* Most recent biopsy positive for prostate cancer
* Currently on or starting active surveillance
* Ability to read, write, and understand English
* BMI >24 kg/m2
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Scheduled to undergo a prostate biopsy in 6 months as part of standard of care for their prostate cancer
* Age > 18 years

Exclusion Criteria:

* Already consuming a severely carbohydrate-restricted (i.e. <20g total carbohydrates per day) or vegetarian diet
* Medical comorbidities that in the opinion of the investigator limits the patient's ability to complete this study
* Anticipate needing prostate cancer therapy within the next 12 months (i.e. surgery, radiation, or hormonal therapy)
* Loss of >10% of body weight within the previous 6 months
* Currently receiving any oral hormonal therapy for prostate cancer or BPH (finasteride, dutasteride, bicalutamide)
* If prior oral hormonal therapy use for prostate cancer or BPH (as defined above), must not have been taking at time of prior biopsy and must be off for at least 3 months prior to study enrollment (oral medications)
* Having ever received any injection hormonal therapy or investigational vaccine for prostate cancer (LHRH agonist, LHRH antagonists, ProstVax, Provenge)
* Current use of weight loss medications including herbal weight loss supplements or enrolled in a diet/weight loss program

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Mean difference change in proliferative index in prostate cancer patients between carbohydrate restricted diet and non-restricted diet groups from pre-study biopsy (baseline) to 6 months. | 6 months
  Proliferative index is measured by Ki67/apoptosis rate

SECONDARY OUTCOMES:
Mean difference in weight loss before and after intervention between between carbohydrate restricted diet and non-restricted diet groups from baseline to 6 months. | 6 months
Mean difference in absolute risk of progression to AUA intermediate risk from baseline to 6 months. | 6 months
  AUA intermediate risk is PSA > 10ng/ml or grade group ≥ 2 or clinical stage ≥ T2b
Mean difference in quality of life between carbohydrate restricted diet and non-restricted diet from baseline to 6 months; measured using EORTC-QLQ-C30. | 6 months
Mean difference in quality of life between carbohydrate restricted diet and non-restricted diet from baseline to 6 months; measured using IPSS. | 6 months
Mean difference in quality of life between carbohydrate restricted diet and non-restricted diet from baseline to 6 months; measured using FACT-Cog. | 6 months
Mean difference in quality of life between carbohydrate restricted diet and non-restricted diet from baseline to 6 months; measured using PROMIS-fatigue. | 6 months
Mean difference in quality of life between carbohydrate restricted diet and non-restricted diet from baseline to 6 months; measured using FACIT-F. | 6 months
Mean difference in quality of life between carbohydrate restricted diet and non-restricted diet from baseline to 6 months; measured using IIEF-5. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedland, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States